CLINICAL TRIAL: NCT03758196
Title: Efficacy and Safety of Renal Sympathetic Denervation From the Adventitia on Resistant Hypertension.
Brief Title: Renal Sympathetic Denervation From the Adventitia on Resistant Hypertension（RSDARH）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HenanICE201802
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Resistant Hypertension
Keywords: renal sympathetic denervation; resistant hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal sympathetic denervation from the adventitia (Experimental): Renal sympathetic denervation from the adventitia of renal artery and optimized medication regimen
  Interventions: Device: Radiofrequency ablation instruments
- optimized medication regimen (No Intervention): optimized medication regimen

INTERVENTIONS:
Device: Radiofrequency ablation instruments — Renal Sympathetic Denervation from the adventitia of renal artery
  Arms: Renal sympathetic denervation from the adventitia

SUMMARY:
As one of the most common chronic diseases,The adult prevalence of hypertension is approximately 26.4% at present and will rise to 29.2% by 2025.Renal sympathetic denervation from the intima of renal artery has emerged as a potential treatment for resistant hypertension. However, renal sympathetic nerve are mainly located in the adventitia,and there is no report on renal sympathetic denervation from the adventitia of renal artery.This study is a multicenter,randomized,single-blind study,and aimed to observe the safety and efficacy of radiofrequency ablation of the renal artery from the adventitia on the basis of laparoscopic techniques for patients with resistant hypertension.

DETAILED DESCRIPTION:
This study is a multicenter,randomized,single-blind study,and aimed to observe the safety and efficacy of radiofrequency ablation of the renal artery from the adventitia on the basis of laparoscopic techniques for patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

1.18 years old ≤ age ≤ 65 years old; 2.Patients with clear diagnosis of resistant hypertension prior to enrollment：On the basis of improving lifestyle, a reasonable and tolerable amount of 3 or more kinds of antihypertensive drugs (including diuretics) for more than one month, clinic SBP≥140mmHg or (and) DBP≥90mmHg, 24 hours dynamic Blood pressure monitoring SBP>130mmHg or (and) DBP>80mmHg; 3.Estimated GFR (eGFR) ≥ 60ml/min/1.73m2; 4.The patient or his legal guardian has signed the informed consent; 5.Patients who are willing and able to perform follow-up visits.

Exclusion Criteria:

1. Patients with secondary hypertension caused by any known cause;
2. pregnant or planning to be pregnant;
3. Patients with renal artery diameter <4mm or length <20mm;
4. Patients with renal artery abnormalities include: hemodynamic or anatomically significant stenosis (≥50%) of renal arteries on either side;renal arterial balloon angioplasty or stenting;renal involvement on either side Multiple renal arteries,and renal arteries supply <75% of the kidneys;abnormal renal artery anatomy,such as tumor expansion;
5. Patients with cardiovascular instability factors includes:acute myocardial infarction within six months,unstable angina or cerebrovascular disease;heart valve disease with significantly altered hemodynamics;
6. Patients with other serious organic diseases;
7. Patients participated in other studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour average systolic blood pressure by ABPM in 6 months after discharge . | Baseline to 6 months

SECONDARY OUTCOMES:
Change in types and doses of antihypertensive medications in 1,3,6,12 months after discharge. | Baseline to 1 months,3 months,6 months,12 months
Change in 24-hour average diastolic blood pressure,daytime and nighttime systolic/diastolic blood pressure by ABPM in 6 months after discharge | Baseline to 6 months
Change in 24-hour average blood pressure,daytime and nighttime systolic/diastolic blood pressure by ABPM in 1,3,12 months after discharge | Baseline to 1 months,3 months,12 months
Change in office systolic/diastolic blood pressure in 1,3,6,12 months after discharge | Baseline to 1 months,3 months,6 months,12 months
Change in systolic/diastolic blood pressure by home blood pressure monitoring in 1,3,6,12 months after discharge | Baseline to 1 months,3 months,6 months,12 months
renal function in 1,3,6,12 months after discharge | Baseline to 1 months,3 months,6 months,12 months
The surgical complications of renal artery perforation,such as stenosis,and dissection associated with radiofrequency surgery.And major cardiovascular and cerebrovascular events ,including cardiac death,stroke and nonfatal- myocardial infarction. | Baseline to 6 months,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chuanyu Gao, Dr., Principal Investigator — Henan Provincial People's Hospital; Jiguang Huang, Dr., Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine;Shanghai Institute of Hypertension
Locations (1):
- Zhengzhou university People's Hospital, Zhengzhou, Henan, China